CLINICAL TRIAL: NCT03623035
Title: Pilot Study on Pain and Sensation After Regional Anesthesia for Total Hip Arthroplasty
Brief Title: Pain and Sensation After Regional Anesthesia - Pilot Study
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00052579
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Results first posted 2019-06-05 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia, Conduction; Osteoarthritis, Hip
Keywords: Lumbar Plexus block; total hip arthroplasty; Arthroplasty, direct anterior approach; Pain
MeSH Terms: conditions — Osteoarthritis, Hip; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lumbar Plexus block Group: This group includes participants that received Lumbar Plexus blocks (LPB) as the regional analgesic technique in a direct anterior approach (DAA) Total Hip Arthroplasty.

SUMMARY:
This study aims to determine spinal resolution and pain levels after the placement of a lumbar plexus block (LPB) and spinal for total hip replacement procedure. This is a pilot study that looks to collect information in order to design a larger, more significant study comparing Quadratus Lumborum blocks (QLB) and Lumbar Plexus blocks.

DETAILED DESCRIPTION:
The Quadratus Lumborum block (QLB) is a newer regional analgesic technique that may be as effective as Lumbar Plexus blocks (LPB) at providing pain control following direct anterior approach (DAA) hip arthroplasty. The purpose of this study is to collect pilot data to help the design of a future randomized study, comparing a QLB to a LPB for DAA procedures. The investigators will assess for spinal resolution below the level of L5/S1 by assessing the presence of pin prick sensation at these levels. This will help determine if pain scores collected at 6hrs reflect analgesia provided by the preoperative LPB alone or if the data is confounded by the presence of spinal anesthesia. This data will help us determine if 6hrs is a feasible primary endpoint to assess pain scores. Additionally, assuming that spinal regression is complete by 6hrs, the VAS pain scores obtained will then be used to perform a power analysis to determine the necessary study size when comparing QLB to LPB for DAA hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have elective total hip arthroplasty with DAA at Davie Medical Center.

Exclusion Criteria:

* Patients will be excluded if they do not receive a lumbar plexus block and spinal anesthesia.
* and/or if they have peripheral neuropathy affecting their feet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Total Hip Arthroplasty surgeries at Davie Medical Center of Wake Forest Baptist Health.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Edwards, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Davie Medical Center, Bermuda Run, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laupacis A, Bourne R, Rorabeck C, Feeny D, Wong C, Tugwell P, Leslie K, Bullas R. The effect of elective total hip replacement on health-related quality of life. J Bone Joint Surg Am. 1993 Nov;75(11):1619-26. doi: 10.2106/00004623-199311000-00006. PMID 8245054
- [Background] Zhao HY, Kang PD, Xia YY, Shi XJ, Nie Y, Pei FX. Comparison of Early Functional Recovery After Total Hip Arthroplasty Using a Direct Anterior or Posterolateral Approach: A Randomized Controlled Trial. J Arthroplasty. 2017 Nov;32(11):3421-3428. doi: 10.1016/j.arth.2017.05.056. Epub 2017 Jun 8. PMID 28662957
- [Background] Capdevila X, Macaire P, Dadure C, Choquet O, Biboulet P, Ryckwaert Y, D'Athis F. Continuous psoas compartment block for postoperative analgesia after total hip arthroplasty: new landmarks, technical guidelines, and clinical evaluation. Anesth Analg. 2002 Jun;94(6):1606-13, table of contents. doi: 10.1097/00000539-200206000-00045. PMID 12032037
- [Background] Post ZD, Orozco F, Diaz-Ledezma C, Hozack WJ, Ong A. Direct anterior approach for total hip arthroplasty: indications, technique, and results. J Am Acad Orthop Surg. 2014 Sep;22(9):595-603. doi: 10.5435/JAAOS-22-09-595. PMID 25157041
- [Background] Williams BA, Kentor ML, Vogt MT, Vogt WB, Coley KC, Williams JP, Roberts MS, Chelly JE, Harner CD, Fu FH. Economics of nerve block pain management after anterior cruciate ligament reconstruction: potential hospital cost savings via associated postanesthesia care unit bypass and same-day discharge. Anesthesiology. 2004 Mar;100(3):697-706. doi: 10.1097/00000542-200403000-00034. PMID 15108988

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumbar Plexus Block Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lumbar Plexus Block Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient Pain Score With Activity
Description: Pain scores will be measured on a verbal pain score when participant sits up in bed. Totals Score range 0-10. Lower scores denote better outcomes.
Time Frame: 6 Hours post block placement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lumbar Plexus Block Group
Number analyzed (Participants) | 10
units on a scale | 1.4 (1.5)

2. Secondary Outcome: Patient Pain Scores at Rest
Description: Pain scores will be measured, when the patient is laying still in bed, on a verbal pain scale. Totals Score range 0-10. Lower scores denote better outcomes.
Time Frame: 6 Hours post block placement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lumbar Plexus Block Group
Number analyzed (Participants) | 10
units on a scale | 1 (1.1)

3. Secondary Outcome: Number of Participants Reporting Pin Prick Sensation
Description: Assessment for spinal resolution below the level of L5/S1 by assessing the presence of pin prick sensation at these levels.
Time Frame: 6 Hours post block placement
Population: Number of patients who had pin prick sensation at the level of L5/S1 6 hours after nerve block and spinal placement.
Measure: Count of Participants; unit: Participants
Arm/Group | Lumbar Plexus Block Group
Number analyzed (Participants) | 10
Participants | 9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 30 days after the day of surgery for each patient.
Description: No patients experienced adverse events.
Arm/Group | Lumbar Plexus Block Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT03623035/Prot_001.pdf